CLINICAL TRIAL: NCT05362721
Title: Assessment of the Impact of Transcatheter Stenting of Aortic Coarctation on the Left Ventricular Afterload and Work Using Left Ventricular Pressure Volume Loops
Brief Title: PV Loop & Coarctation Study
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2019-27404
Record Dates: First submitted 2022-04-15; First posted 2022-05-05 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Coarctation of Aorta
Keywords: Coarctation of Aorta; COA
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pressure-volume loop catheter
  Interventions: Diagnostic Test: Pressure-volume loop catheter

INTERVENTIONS:
Diagnostic Test: Pressure-volume loop catheter — The cardiac catheterization procedure will be done according to standard protocol as part of the standard clinical care. This has become the standard of care in any patient in which it feasible and is performed with low risk.

SUMMARY:
Coarctation of the aorta accounts for 4-7% of all congenital heart disease. While stent therapy, when feasible, is the standard of care for coarctation, it may not completely improve the work (and afterload) of the heart due to its effects on the elasticity of the aorta. This study will provide the information needed to understand the effects of current management on the cardiac mechanics and work.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 years of age and older and adults of all races and both sexes referred for elective cardiac catheterization and stent therapy for coarctation
* Those who provide informed consent for study participant.

Exclusion Criteria:

* Children who undergo other interventions in addition to the coarctation
* Children with single ventricle physiology.
* Renal impairment
* Participant unwilling to sign a consent form.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for elective cardiac catheterization and stent therapy for coarctation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular afterload measured by arterial elastance | Immediately following intervention
  Arterial elastance (Ea) is measured by the pressure volume (PV) loop catheter in the left ventricle. The PV loop catheter measures pressure and volume simultaneously during the entire cardiac cycle. Arterial elastance is a measure of ventricular afterload and will be calculated using previously described formula;
  Ea (arterial elastance): Ea = Pend systole/ SV
  (where P, is pressure at end systole, and SV is stroke volume).
  Elastance will be reported as a continuous variable in mmHg/mL with a higher number indicating an increase in elastance and a negative number indicating a decrease in elastance. Change in elastance before and after stent placement will be compared using paired T test.

SECONDARY OUTCOMES:
Change in left ventricular performance measured by ESPVR | Immediately following intervention
  The end systolic pressure volume relationship (ESPVR) summarizes ventricular systolic function and is measured as a slope of End systolic ventricular elastance (Ees) and volume-axis intercept Vo such that ESP = Ees (ESV-Vo) (ESP = end-systolic pressure, ESV = end-systolic volume, Vo represents the unstressed volume, which is the volume required to fill the ventricle before pressure rises). Shifts of the ESPVR occur with changes in ventricular contractility such that increases in contractility are associated with upward/leftward shifts of the ESPVR. ESPVR is obtained by analysing the data and PV loops obtained by PV loop catheter in the left ventricle before and after intervention. It will be depicted as a continuous variable in mmHg/ml as well as graphically as a slope. Changes before and after intervention will be compared as shifts in ESPVR.
Change in left ventricular work as measured by Stroke Work | Immediately following intervention
  Stroke work (SW) is a continuous variable that measures the work done by the left ventricle in ejecting blood in one cardiac cycle. It is the area under one loop and is measured in mmHg.ml. SW is obtained by analysing the data and PV loops obtained by PV loop catheter in the left ventricle before and after intervention. SW before and after intervention will be compared as continuous variables using appropriate statistical tests.
Change in left ventricular efficiency as measured by ventricular arterial coupling | Immediately following intervention
  VA coupling is calculated by the ratio of effective arterial elastance (Ea), a measure of afterload, to LV endsystolic elastance (Ees), a relatively load independent measure of LV chamber performance. Both these measures are expressed in mmHg/ml and as continuous variables. Normal determined Ea and Ees values in resting subjects are 2.2 ± 0.8 mmHg/ml and 2.3 ± 1.0 mmHg/ml, respectively. When Ea/Ees ratio is approximately equal to 1.0, LV and arterial system are optimally coupled to produce stroke work, a measure of the efficiency of LV work, corresponding to the product of systolic arterial pressure and stroke volume, and related to oxygen consumption. When Ea/Ees ratio is <1.0, the stroke work remains close to optimal values, but when EA/EES ratio is >1.0, the stroke work significantly falls, and the LV becomes progressively less efficient. We will compare VA coupling before and after intervention and will be analyzed as continuous variables with appropriate statistical tests.

CONTACTS AND LOCATIONS:
Overall Officials: Gurumurthy Hiremath, Principal Investigator — University of Minnesota
Locations (7):
- United States (7):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital of Boston, Boston, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas-Southwestern, Dallas, Texas